CLINICAL TRIAL: NCT06088680
Title: A Post Market Multicentre Retrospective Study of Glycar Bovine Pericardial Patch With AldeCaptm Technology (Aka SJM With EnCaptm Technology) in Cardiac and Vascular Repair or Reconstruction Surgery (CIP-003)
Brief Title: Post Market Observational Retrospective Study of Glycar Bovine Pericardial Patch (CIP-003)
Status: Completed | Type: Observational
Sponsor: GLYCAR SA (Pty) Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-003
Record Dates: First submitted 2023-10-02; First posted 2023-10-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Defect; Cardiac Anomaly; Pericardial Defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open Label- Glycar Pericardial Patch: patients undergoing cardiovascular repair or reconstruction surgery under standard clinical care with the commercially available Glycar Pericardial Patch.
  Interventions: Device: Glycar Pericardial Patch

INTERVENTIONS:
Device: Glycar Pericardial Patch — Glycar Bovine pericardial patch with AldeCaptm Technology (aka SJM with EnCaptm technology)

SUMMARY:
The overall purpose of this observational Post Market Clinical Follow Up (PMCF) study is to ensure continued acceptability of the benefit risk ratio by assessment of safety and performance, in patients undergoing cardiovascular repair or reconstruction surgery under standard clinical care with the commercially available Glycar Pericardial Patch.

DETAILED DESCRIPTION:
To comply with Medical Device Regulation (MDR) Post Market Clinical Follow Up (PMCF) requirements through proactive ongoing assessment of the safety, efficacy, and performance of the commercially available Glycar Pericardial Patch in patients undergoing cardiovascular repair or reconstruction surgery.

This real-world evidence retrospective data collection single-arm multicentre, observational, non-interventional study will enrol up to a minimum of 50 consecutive participants who meet inclusion criteria, in 2-3 centres. The study is aimed at providing real-world evidence of the Glycar Pericardial patch.

Retrospective data analysis will include collected clinical data from consecutive participants with a minimum of 2 years follow up, meaning from 30 June 2020 and going back in time. The quality of medical history being recorded is believed to be more reliable and complete in the most recent years. Therefore, it was decided to start enrolling consecutive participants in a reverse chronological order.

ELIGIBILITY:
Inclusion Criteria:

* If no waiver has been granted by the Ethics committee: Participants (all age) or legal guardian has signed the informed consent
* Participant has undergone a cardiac or vascular procedure which falls within the indications for use and required the use of Glycar Pericardial Patch

Exclusion Criteria:

- There are no study specific exclusion criteria. Participants have already been treated per standard clinical practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing cardiovascular repair or reconstruction surgery under standard clinical care with the commercially available Glycar Pericardial Patch.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Reintervention | Within < 30 days post procedure
  Incidence of patch related reintervention
Mortality | Within < 30 days post procedure
  Incidence of patch related mortality

SECONDARY OUTCOMES:
Reintervention | Up to 2 years
  Incidence of patch related reintervention
Mortality | Up to 2 years
  Incidence of patch related mortality
Infection | Up to 2 years
  Rate of occurrence of Patch infection (such as endocarditis)
Thrombus formation | Within < 30 days post procedure
  Incidence of thrombus formation
Unplanned reoperations | Up to 2 years
  The total number of unplanned reoperations required in patients over the FU period which include the repair or alteration of the surgical area around the patch. Patients with planned reoperations at the time of the primary index procedure will not be considered
Unanticipated AEs | Up to 2 years
  Incidence of patch Unanticipated Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Red Cross War Memorial Children's Hospital, Cape Town, Rondebosch, South Africa

IPD SHARING:
Plan to Share IPD: No